CLINICAL TRIAL: NCT03566992
Title: Effect of Location of Feeding on Glycemic Control in Critically Ill Patients (ELF)
Acronym: ELF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Winchester Medical Center (Other)
Collaborators: Halyard Health (Industry)
Responsible Party: Principal Investigator, Padmaraj Duvvuri, Principal Investigator, Critical Care Physician, Winchester Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WinchesterMC
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Glucose Metabolism Disorders; Critical Illness
MeSH Terms: conditions — Glucose Metabolism Disorders; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric Tube Placement (Active Comparator): Nasoenteric tube placed in the stomach.
  Interventions: Procedure: Gastric
- Small bowel (Experimental): Nasoenteric tube placed in the small bowel.
  Interventions: Procedure: Gastric

INTERVENTIONS:
Procedure: Gastric — Placement of a nasoenteric tube

SUMMARY:
The purpose of this study is to investigate the effect of location of feeding on glycemic control in critically ill patients.

The investigators hypothesize that glycemic control in critically ill patients who receive enteral nutrition through postpyloric location (beyond stomach) will have better glycemic control compared to critically ill patients fed gastrically.

DETAILED DESCRIPTION:
Randomization will happen after initial stabilization phase which may last up to 24 hours till when patient may or may not have an enteric access. If enteral access is gained and patient is screened in for the study using inclusion and exclusion criteria, a consent shall be obtained for enrollment. The tube may be continued to be used if randomized in group A. If patient is randomized to group B, a postpyloric placement will be achieved.

Randomization using computer software and a unique identification number will be assigned to every intubated patients who may need mechanical ventilation or tube feed for more than 48 hours.

Randomization will be considered incomplete and the case will be excluded if the process of assigning group, confirmation of placement of appropriate group specific tube and nutrition is not initiated within 24 hours.

If patient is randomized into group A, a bedside RN or the intensivist will place a Salem Sump gastric tube. A nutrition consult for tube feed will be obtained. Confirmation of gastric placement and not a postpyloric placement will be based on the length of the orogastric/nasogastric tube and a standard chest radiograph obtained routinely after intubation. The NG or OG tube should not be more than 65 cm in most cases to prevent it from migrating into the postpyloric location. A standard enteral tube feed formula will be initiated. Blood sugars checked via basic metabolic (at least daily) panel and point-of-care glucose tests (at least every 6 hours) will be obtained. Data collection and Salem Sump placement will be confirmed by the studying team and will not be known to the RD prescribing the nutrition.

If a patient is randomized into group B, a trained RN or RD will place the small-bore feeding feeding tube in the postpyloric position. The effort will be to assure jejunal placement, but postpyloric placement should be sufficient. If for some reason, the small-bore tube cannot be passed beyond pylorus, then sufficient length will be left in IRB the stomach and the case will be noted to have not had the postpyloric placement.

A per protocol analysis and an intention to treat analysis will be carried in the end to take into consideration cases when placement of tube in certain location could not be achieved.

If a feeding tube becomes occluded, it will be replaced with a new tube within 12 hours. If the patient had a postpyloric tube and the new tube cannot be positioned in the postpyloric location, the patient's involvement in the study will be halted (no further data collection).

A standard enteral tube feed formula will be initiated. Blood sugars checked via basic metabolic (at least daily) panel and point-of-care glucose tests (at least every 6 hours) will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18 years or above) patients admitted in the critical care unit on mechanical ventilation for at least 48 hours
2. Orders for tube feeding

Exclusion Criteria:

1. Intubated for less than 48 hours (suspected insufficient time for the role of feeding mode to affect glycemic control)
2. Patients not being fed (such as DKA, GI bleed, obstruction, ileus, etc)
3. Pre-existing PEG/PEJ tubes
4. Surgically altered upper and middle GI tract such as partial gastrectomy, gastric bypass surgeries etc. (patients with ileostomy and colostomy may still be included if the enteral route is used for nutrition)
5. No informed consent
6. Primary attending finds medical necessity to have a specific type of tube preventing randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Nasoenteric tube placement | Intubated patients >48 hours and up to 7 days.
  Investigate the effect of location of feeding on glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: Padmaraj Duvvuri, MD, Study Director — Winchester Medical Center
Locations (1):
- Winchester Medical Center, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Metheny NA, Clouse RE, Chang YH, Stewart BJ, Oliver DA, Kollef MH. Tracheobronchial aspiration of gastric contents in critically ill tube-fed patients: frequency, outcomes, and risk factors. Crit Care Med. 2006 Apr;34(4):1007-15. doi: 10.1097/01.CCM.0000206106.65220.59. PMID 16484901
- [Background] Di Bartolomeo AE, Chapman MJ, V Zaknic A, Summers MJ, Jones KL, Nguyen NQ, Rayner CK, Horowitz M, Deane AM. Comparative effects on glucose absorption of intragastric and post-pyloric nutrient delivery in the critically ill. Crit Care. 2012 Sep 17;16(5):R167. doi: 10.1186/cc11522. PMID 22985684
- [Background] Pournaras DJ, Aasheim ET, Bueter M, Ahmed AR, Welbourn R, Olbers T, le Roux CW. Effect of bypassing the proximal gut on gut hormones involved with glycemic control and weight loss. Surg Obes Relat Dis. 2012 Jul-Aug;8(4):371-4. doi: 10.1016/j.soard.2012.01.021. Epub 2012 Mar 3. PMID 22480751
- [Background] Luttikhold J, van Norren K, Rijna H, Buijs N, Ankersmit M, Heijboer AC, Gootjes J, Hartmann B, Holst JJ, van Loon LJ, van Leeuwen PA. Jejunal feeding is followed by a greater rise in plasma cholecystokinin, peptide YY, glucagon-like peptide 1, and glucagon-like peptide 2 concentrations compared with gastric feeding in vivo in humans: a randomized trial. Am J Clin Nutr. 2016 Feb;103(2):435-43. doi: 10.3945/ajcn.115.116251. Epub 2016 Jan 13. PMID 26762368